CLINICAL TRIAL: NCT06636708
Title: Evaluation of Nanodropper-mediated Microdrops vs. Standard Drops of 0.5% Proparacaine HCl
Brief Title: Efficacy of Nanodropper-mediated Topical Anesthetic
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Aakriti G. Shukla, Associate Professor of Ophthalmology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Device Feasibility
Other Study IDs: AAAU9824
Record Dates: First submitted 2024-10-08; First posted 2024-10-15 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Corneal Diseases; Effectiveness of Microdrops
Keywords: Corneal anesthesia; Nanodropper
MeSH Terms: conditions — Corneal Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard Eye Drops (Active Comparator): Eyes randomized to this arm will receive a standard drop of 0.5% proparacaine HCl
  Interventions: Combination Product: Standard Eye Drop Bottle with Proparacaine HCl 0.5%
- Nanodropper (Experimental): Eyes randomized to this arm will receive a Nanodropper-mediated microdrop of 0.5% proparacaine HCl
  Interventions: Combination Product: Nanodropper and Proparacaine HCl 0.5%

INTERVENTIONS:
Combination Product: Nanodropper and Proparacaine HCl 0.5% — The Nanodropper is an eyedrop bottle adaptor that creates smaller eyedrops by coupling to an existing eyedrop bottle. This intervention involves the administration of proparacaine HCl 0.5% using the Nanodropper.
  Arms: Nanodropper
Combination Product: Standard Eye Drop Bottle with Proparacaine HCl 0.5% — This intervention involves administration of proparacaine HCl 0.5% using a standard eye drop bottle.
  Arms: Standard Eye Drops

SUMMARY:
The goal of this clinical trial is to compare the onset and duration of numbness of the surface of the eye following the administration of numbing drops, called proparacaine, using either a standard eye drop bottle or a "Nanodropper" adaptor. The Nanodropper is designed to administer smaller-sized drops, or microdrops.

Participants will:

1. Complete a baseline eye exam.
2. Receive a numbing drop using a standard dropper in one eye and the Nanodropper in the other eye.
3. Have their eyes tested for numbness at specific time points (30 seconds, 1, 2, 5, and 10 minutes after getting the drops).
4. Tell the researchers if they feel pain during the eye sensation tests.
5. Complete a survey about their experience with the eyedrops and testing procedure.

This study could help us find a way to use less medication while still effectively administering eye medications, potentially saving money and reducing medical waste.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide informed consent for topical anesthesia delivery
2. Ability to verbally respond to pain
3. At least 18 years of age

Exclusion Criteria:

1. Have a contraindication to local anesthetics
2. History of intravitreal injections
3. History of ocular surgery
4. History of vitreous or retinal surgery
5. Preexisting diagnosis of ocular surface disease requiring punctal plug placement
6. Evidence of any current ocular inflammation
7. Any previous ocular condition (i.e., neurotrophic keratitis, herpetic eye disease, presence of a corneal graft, etc.) that has permanently altered the native sensation of the ocular surface
8. Use of contact lenses in the past 2 weeks
9. Use of exclusionary medications: Topical steroid drops, non-steroidal anti-inflammatory drops, intraocular pressure lowering eye drops, any anti-viral medications used for herpes, opioids

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2024-12-12 (Actual); Primary Completion 2025-04-24 (Actual); Study Completion 2025-04-24 (Actual)

PRIMARY OUTCOMES:
Corneal Anesthesia | 5 minutes
  The primary outcome is the percent or proportion of subjects that achieve anesthesia at the 5-minute time point

CONTACTS AND LOCATIONS:
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] St Peter DM, Steger JS, Patnaik JL, Davis N, Kahook MY, Seibold LK. Reduction of Eyedrop Volume for Topical Ophthalmic Medications with the Nanodropper Bottle Adaptor. Med Devices (Auckl). 2023 Apr 6;16:71-79. doi: 10.2147/MDER.S397654. eCollection 2023. PMID 37056302
- [Background] Palmer DJ, Robin AL, McCabe CM, Chang DF; Ophthalmic Instrument Cleaning and Sterilization Task Force. Reducing topical drug waste in ophthalmic surgery: multisociety position paper. J Cataract Refract Surg. 2022 Sep 1;48(9):1073-1077. doi: 10.1097/j.jcrs.0000000000000975. PMID 35608314
- [Background] Moore DB, Walton C, Moeller KL, Slabaugh MA, Mudumbai RC, Chen PP. Prevalence of self-reported early glaucoma eye drop bottle exhaustion and associated risk factors: a patient survey. BMC Ophthalmol. 2014 Jun 13;14:79. doi: 10.1186/1471-2415-14-79. PMID 24927769